CLINICAL TRIAL: NCT06543940
Title: Pharmacokinetics of Vancomycin in Patients Receiving Continuous Veno-Venous Hemodiafiltration (CVVHDF) with the Absorptive OXiris Membrane
Brief Title: Pharmacokinetics Vancomycin CVVHDF with OXiris Membrane
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Chidtawan Hirunsomboon, lecturer faculty of pharmacy, Mahidol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: MUPY00001
Record Dates: First submitted 2024-07-26; First posted 2024-08-09 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: AKI - Acute Kidney Injury
Keywords: vancomycin; CRRT; oXiris membrane
MeSH Terms: conditions — Acute Kidney Injury | interventions — Vancomycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Vancomycin (Experimental): administration with vancomycin 7.5 to 10 mg/kg IV q 12 hours in patient received CRRT with oXiris membrane
  Interventions: Drug: Vancomycin

INTERVENTIONS:
Drug: Vancomycin — vancomycin dose is 7.5 to 10 mg/kg

SUMMARY:
This study is a general pharmacokinetic investigation of vancomycin in patients receiving continuous veno-venous hemodiafiltration (CRRT) with the oXiris membrane. This membrane offers the added benefit of absorbing inflammatory cytokines. In vitro studies show that vancomycin is reduced by around 20 percent in patients using the AN69ST membrane, which is part of the oXiris membrane's structure. However, there is currently a lack of in vivo studies demonstrating the impact of the oXiris membrane on vancomycin levels. Therefore, the hypothesis of this study is that vancomycin is also reduced by absorption in the oXiris membrane. This study measures the levels of vancomycin in these patients to determine the pharmacokinetic parameters.

DETAILED DESCRIPTION:
This study monitors the levels of the maintenance dose of vancomycin in patients receiving continuous renal replacement therapy (CRRT) with the CVVHDF mode using the oXiris membrane. Blood samples were drawn from the A-line at the following time points: 0 (predose), 2, 3, 4, 5, 6, 8, and 12 hours after drug administration. The area under the curve (AUC) of the drug was calculated using the Phoenix WinNonlin program. Additionally, we reported the pharmacokinetic profile of this drug in patients with acute kidney injury (AKI) undergoing CRRT with the oXiris membrane.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged more than 18 years.
* Admitted to the intensive care unit of Ramathibodi Hospital.
* Under continuous renal replacement therapy (CRRT) with CVVHDF using oXiris filter.
* Received vancomycin at least once after starting CRRT with CVVHDF using oXiris filter.
* who have signed the informed consent document.

Exclusion Criteria:

* Patients with a history of vancomycin allergy.
* Patients expected to die within 24 hours after inclusion in study.
* Patients with circuit clotting occurring more than 2 hours during the blood draw period.
* Patients treated with extracorporeal membrane oxygenation (ECMO).
* Patients with a history of kidney transplantation.
* Pregnant or breastfeeding women.
* Patients who have decided to receive palliative care.
* Patients on hemodialysis or peritoneal dialysis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
AUC of vancomycin | at 0 pre-dose, 2,3,4,5,6,8 and 12 hours after intervention vancomycin
  calculated AUC of vancomycin by 8 points of drug level. (at 0 pre-dose, 2,3,4,5,6,8 and 12 hours after administration)

SECONDARY OUTCOMES:
To determine the Cmax of vancomycin | 1 year
  calculated Cmax of vancomycin in these patient by phoenix winnonlin software.
30-day mortality rate | 30 day after intervention period
  monitor mortality rate at 30 days after received maintenance dose
percentage of patients who, receiving AUC/MIC ratio within the range of 400 to 600 mg*h/L. | 1 years
  calculate percent sample who AUC with in target by number sample in target divide to total population.
incidence of adverse effects of vancomycin | 1 years
  record the incidence of adverse effects during the intervention period.
renal recovery rate at 30 days | 30 day after intervention period
  monitor renal replacement therapy status at 30 days after received maintenance dose
To determine the elimination rate constant (Ke) of vancomycin | 1 years
  calculated Ke of vancomycin in these patient by phoenix winnonlin software.
To determine the volume of distribution (Vd) of vancomycin | 1 years
  calculated Vd of vancomycin in these patient by phoenix winnonlin software.
To determine the half life of vancomycin | 1 years
  calculated half life of vancomycin in these patient by phoenix winnonlin software.

CONTACTS AND LOCATIONS:
Locations (1):
- Facullty of Pharmacy Mahidol University, Bangkok, Payathi, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bruniera FR, Ferreira FM, Saviolli LR, Bacci MR, Feder D, da Luz Goncalves Pedreira M, Sorgini Peterlini MA, Azzalis LA, Campos Junqueira VB, Fonseca FL. The use of vancomycin with its therapeutic and adverse effects: a review. Eur Rev Med Pharmacol Sci. 2015 Feb;19(4):694-700. PMID 25753888
- [Background] Rybak MJ, Le J, Lodise TP, Levine DP, Bradley JS, Liu C, Mueller BA, Pai MP, Wong-Beringer A, Rotschafer JC, Rodvold KA, Maples HD, Lomaestro BM. Therapeutic monitoring of vancomycin for serious methicillin-resistant Staphylococcus aureus infections: A revised consensus guideline and review by the American Society of Health-System Pharmacists, the Infectious Diseases Society of America, the Pediatric Infectious Diseases Society, and the Society of Infectious Diseases Pharmacists. Am J Health Syst Pharm. 2020 May 19;77(11):835-864. doi: 10.1093/ajhp/zxaa036. No abstract available. PMID 32191793
- [Background] DelDot ME, Lipman J, Tett SE. Vancomycin pharmacokinetics in critically ill patients receiving continuous venovenous haemodiafiltration. Br J Clin Pharmacol. 2004 Sep;58(3):259-68. doi: 10.1111/j.1365-2125.2004.02143.x. PMID 15327585
- [Background] Chaijamorn W, Jitsurong A, Wiwattanawongsa K, Wanakamanee U, Dandecha P. Vancomycin clearance during continuous venovenous haemofiltration in critically ill patients. Int J Antimicrob Agents. 2011 Aug;38(2):152-6. doi: 10.1016/j.ijantimicag.2011.04.010. Epub 2011 Jun 1. PMID 21636256
- [Background] Onichimowski D, Nosek K, Ziolkowski H, Jaroszewski J, Pawlos A, Czuczwar M. Adsorption of vancomycin, gentamycin, ciprofloxacin and tygecycline on the filters in continuous renal replacement therapy circuits: in full blood in vitro study. J Artif Organs. 2021 Mar;24(1):65-73. doi: 10.1007/s10047-020-01214-8. Epub 2020 Oct 8. PMID 33033945